CLINICAL TRIAL: NCT07144891
Title: Sperm DNA Fragmentation Among Other Variableas a Predictor for Outcome After Varicocelectomy,
Brief Title: sperDNA Fragmentation a a Predictor for Outcome After Varicocelectomy,m
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Deif Abdelghani Ghidan, Principal Investigator, Assiut University
Other Study IDs: SDV
Record Dates: First submitted 2025-05-05; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: DNA Damage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1
  Interventions: Genetic: Sperm DNA fragmentation

INTERVENTIONS:
Genetic: Sperm DNA fragmentation — Estimation of sperm DFI level with sperm chromatin dispersion

SUMMARY:
Varicocele is often associated with infertility and reduction in sperm quality, and it is one of the most common causes of reversible male infertility.

The exact mechanism of infertility caused due to varicocele formation remains unclear. One of the suggested theories is related to increased oxidative stress that causes sperm DNA damage, including DNA fragmentation, and is correlated with the decreased capacity of spermatozoa to fertilize oocytes during normal fertilization and assisted reproduction techniques. This is supported by the evidence that there is a higher prevalence of DNA fragmentation in varicocele patients and a correlation between the presence of varicocele and impaired sperm DNA integrity.

Several tests have been developed to better assess the fertility potential of sperm, including those designed to measure sperm deoxyribonucleic acid (DNA) fragmentation (SDF). The sperm DNA fragmentation index (DFI) is a potential parameter for fertility investigation, reflecting sperm DNA integrity and damage.

DETAILED DESCRIPTION:
Varicocele is often associated with infertility and reduction in sperm quality, and it is one of the most common causes of reversible male infertility.

The prevalence of clinically relevant varicocele ranges from 5 to 20%. It has affected 19-41% of men with primary infertility and 45-81% of men with secondary infertility.

The exact mechanism of infertility caused due to varicocele formation remains unclear. One of the suggested theories is related to increased oxidative stress that causes sperm DNA damage, including DNA fragmentation, and is correlated with the decreased capacity of spermatozoa to fertilize oocytes during normal fertilization and assisted reproduction techniques. This is supported by the evidence that there is a higher prevalence of DNA fragmentation in varicocele patients and a correlation between the presence of varicocele and impaired sperm DNA integrity.

Several tests have been developed to better assess the fertility potential of sperm, including those designed to measure sperm deoxyribonucleic acid (DNA) fragmentation (SDF). The sperm DNA fragmentation index (DFI) is a potential parameter for fertility investigation, reflecting sperm DNA integrity and damage.

Current guidelines recommend that varicoceles be treated in cases of documented infertility, palpable varicocele, normal or potentially corrected female fertility, and at least one abnormal sperm parameter with no clear statement about abnormal sperm DNA or function Furthermore, Zavattaro et al. reported that around 15% of varicocele patients with normal semen analysis are diagnosed as infertile .

Due to conflicting studies and a lack of high-quality evidence, it is unclear how SDF testing should best be applied in the evaluation and treatment of infertile men, making SDF an active area of research [. Although most men with abnormal semen parameters will have an improvement in semen parameters after varicocelectomy, until recently we had no way to accurately predict which men would respond positively to VC repair .

While preoperative total motile sperm count (TMSC) coupled with sperm concentration can be a significant predictor of semen improvement and pregnancy after varicocelectomy , Despite the presence of numerous studies about the prognostic variables with VC repair, little well designed studies were published about the role of more objective factors as sperm DNA damage and oxidative stress as a prognostic factors with VC repair in infertile men. These variables were found to be more objective predictors for normal and assisted conception even more than conventional semen parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been diagnosed with VC (GII and GIII) by physical examination and scrotal color Doppler ultrasonography.
* Patients with stable relationships.
* In the control group, those with high SDF.
* Patients with documented infertility.
* Normal female partners or having correctable cause of infertility.
* Patients age from 20 to 45 years old.

Exclusion Criteria:

Patients with a history of scrotal and spermatic cord injuries and congenital genitourinary abnormalities.

* Patients with systemic or endocrine disease, cryptorchidism, hypogonadism, genital infection, hormonal treatment and azoospermic patients.
* Recurrent varicocele.
* Patients with any other disease that may cause VC (such as external kidney tumor, hydronephrosis, etc.)
* Smoker patients and others risk factors (x ray, nuclear) workers
* Abnormal or uncorrectable female factor. 7- Single patient.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: infertile male from 20 years old to 45 years old
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
we will assess sperm DNA fragmentation as a pridector for outcome of varicoelectomy in a group of infertile males with palpable varicocele. | 1 year
  In this study, we will assess sperm DNA fragmentation index as a pridector for outcome of varicoelectomy in a group of infertile males with palpable varicocele.

REFERENCES:
- [Background] Birowo P, Rahendra Wijaya J, Atmoko W, Rasyid N. The effects of varicocelectomy on the DNA fragmentation index and other sperm parameters: a meta-analysis. Basic Clin Androl. 2020 Sep 10;30:15. doi: 10.1186/s12610-020-00112-6. eCollection 2020. PMID 32944248
- [Background] Wang L, Zheng L, Jiang H, Jiang T. Does Sperm DNA Fragmentation Index Continuously Decrease Over Time After Varicocelectomy in Varicocele-Induced Infertility? A Systematic Review and Meta-Analysis. Am J Mens Health. 2024 Sep-Oct;18(5):15579883241285670. doi: 10.1177/15579883241285670. PMID 39376021
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC7488296/
- Available data/document: article — https://pmc.ncbi.nlm.nih.gov/articles/PMC7488296/